CLINICAL TRIAL: NCT01238302
Title: Arthroscopic Rotator Cuff Repair With Platelet-Rich Plasma(PRP) in Large to Massive Tears : A Randomized Controlled Trial
Brief Title: Arthroscopic Rotator Cuff Repair With Platelet-Rich Plasma(PRP) in Large to Massive Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunchul Jo, Assistant Professor, SMG-SNU Boramae Medical Center., Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRM-10-03
Record Dates: First submitted 2010-11-08; First posted 2010-11-10 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional group (Placebo Comparator)
  Interventions: Procedure: Conventional arthroscopic rotator cuff repair
- PRP group (Experimental)
  Interventions: Procedure: Arthroscopic rotator cuff repair with PRP

INTERVENTIONS:
Procedure: Conventional arthroscopic rotator cuff repair — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4-5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repair of full thickness rotator cuff tear was done with suture anchors.
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  Arms: Conventional group
Procedure: Arthroscopic rotator cuff repair with PRP — * Under general anesthesia, the patient was placed in the lazy lateral decubitus position on the operating table.
  * The surgical area was prepared and draped with Betadine.
  * Small stab incisions were made in the creation of 4-5 portals as needed.
  * A scope was explored via the arthroscopic portal into the GH joint & subacromial space.
  * Repair of full thickness rotator cuff tear was done with suture anchors.
  * After tying sutures of the medial row, PRP gels were applied on the repair site.
  * The lateral row was secured using suture anchors.
  * The skin was closed with Nylon or medical staples.
  * Sterile dressing was applied on surgical wound.
  Arms: PRP group

SUMMARY:
* The purpose of this study is to compare the clinical and anatomical outcomes of rotator cuff repair with Platelet-Rich Plasma(PRP) and conventional rotator cuff repair in treatment of large to massive rotator cuff tears.
* PRP application to arthroscopic rotator cuff repair would accelerate recovery after arthroscopic rotator cuff repair in terms of pain relief, functional outcomes, overall satisfaction, and enhance structural integrity of repaired tendon.

ELIGIBILITY:
Inclusion Criteria:

large to massive rotator cuff tear as a determined by clinical examination and MR prior to surgery.

Exclusion Criteria:

* previous history of shoulder surgery
* acute trauma
* chronic dislocation
* pyogenic infection
* rotator cuff arthropathy with glenohumeral osteoarthritis and superior migration of the humeral head
* showed abnormal serological test results
* thrombocytopenia (platelets less than 15000 per microliter)
* had been received anti-platelet medication
* psychiatric problems that precludes informed consent or inability to read or write
* other serious problems that preclude participation of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
structural integrity of repaired rotator cuff tendon | postoperative 9months
  To evaluate structural outcomes, magnetic resonance(MR)imaging or computed tomography arthrography were used at minimum postoperative 9months.
  The structural integrity was evaluated using Sugaya's method;
  * type I, sufficient thickness with homogenously low intensity
  * type II, insufficient thickness partial high intensity
  * type III, insufficient thickness without discontinuity (thinned cuff)
  * type IV, presence of minor discontinuity
  * type V, presence of a major discontinuity
  Type I, II, and III were considered as healed, while type IV, and V were considered as retear.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hyunchul Jo, M.D., Ph.D, Principal Investigator — Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, South Korea